CLINICAL TRIAL: NCT03203642
Title: A Double-blind Randomized Parallel Group Study of the Efficacy and Safety of Tesevatinib in Subjects With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Study of the Efficacy and Safety of Tesevatinib in Subjects With ADPKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17675; KD019-211 (Other: Kadmon)
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Autosomal Dominant Polycystic Kidney; ADPKD
Keywords: ADPKD; Autosomal Dominant Polycystic Kidney Disease; Polycystic Kidney; Tesevatinib; Polycystic Kidney Disease; PKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases | interventions — XL647

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tesevatinib (Experimental): Participants received tesevatinib 50 mg tablet orally once daily (QD) for up to 25.3 months.
  Interventions: Drug: Tesevatinib
- Placebo (Placebo Comparator): Participants received placebo matched to tesevatinib tablet orally QD for up to 25.3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tesevatinib — Pharmaceutical form: Tablet; Route of administration: orally
  Other Names: KD019
  Arms: Tesevatinib
Drug: Placebo — Pharmaceutical form: Tablet (identical to tesevatinib); Route of administration: orally
  Arms: Placebo

SUMMARY:
The goal of the study was to compare and evaluate safety and efficacy of tesevatinib 50 milligrams (mg) versus placebo in participants with autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
Safety and efficacy of 50 mg tesevatinib in comparison to placebo in participants with ADPKD was assessed.

The primary purpose of this study was focused on evaluating the change from Baseline in height-adjusted total kidney volume (htTKV) as measured by magnetic resonance imaging (MRI) at Months 12, 18, and 24, and 30 days post-dose in participants with ADPKD treated with tesevatinib or placebo.

If eligible for the study participation, participants were randomly assigned to either investigational treatment group or placebo group. Treatment group received 50 mg tesevatinib once daily for 24 months and control group received the placebo once daily for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD diagnosis based on Ravine's criteria.
* Cysts of at least 1 centimeter.
* Estimated glomerular filtration rate greater than or equal to (>=) 25 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) and less than or equal to (<=) 90 mL/min/1.73 m^2, using the Modification of Diet in Renal Disease-4 variable formula.
* htTKV must meet the following requirements: >= 500 milliliters (mL) for participants 18-35 years of age; >= 750 mL for participants 36-49 years of age; >= 900 mL for participants 50-60 years of age.
* The participant had the following laboratory values:

Platelets greater than (>) lower limit of normal (LLN); Hemoglobin > 9 grams per deciliter; Total bilirubin <= 1.5 milligrams per deciliter; Aspartate aminotransferase less than (<) 2.5*upper limit of normal (ULN); Alanine aminotransferase < 2.5*ULN; Prothrombin time/partial thromboplastin time <=1.5*ULN; Serum potassium levels within normal limits; Serum magnesium levels within normal limits; Albumin >= LLN; Amylase <=1.5*ULN; Lipase <=1.5*ULN; Prothrombin time and partial thromboplastin time <=1.5*ULN; International normalized ratio (INR) <=1.5, except those participants taking warfarin who must have INR <=3.

* Female participants of childbearing potential with negative pregnancy test at screening.
* If sexually active, the participant agreed to use 2 accepted methods of contraception during the course of the study and for 6 months after their last dose of study drug.

Exclusion Criteria:

* Previous nephrectomy.
* Kidney transplant.
* Tuberous sclerosis.
* Hippel-Lindau disease.
* Acquired cystic disease.
* Congenital absence of 1 kidney and/or need for dialysis or transplantation in the foreseeable future.
* Moderate hematuria.
* Uncontrolled hypertension.
* Presence of renal or hepatic calculi (stones) causing symptoms.
* Received any investigational therapy within 30 days prior to initiation of therapy (Day 1 visit).
* Received tolvaptan 30 days prior to initiation of therapy (Day 1 visit).
* Received active treatment for urinary tract infection 4 weeks prior to initiation of therapy (Day 1 visit).
* History of pancreatitis or known risk of pancreatitis.
* The participant met any of the following cardiac criteria:
* Mean QTc interval corrected for heart rate using Fridericia's formula (QTcF) of >450 milliseconds.
* History of torsade de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 50 beats per minute), heart block (excluding first-degree block, being PR interval prolongation only), congenital long QT syndrome or new ST segment elevation or depression or new Q wave on electrocardiogram.
* Participants with a history of atrial arrhythmias were discussed with the Medical Monitor.
* Family history of congenital long QT syndrome or unexplained cardiac death.
* Symptomatic heart failure (per New York Heart Association guidelines), unstable angina, myocardial infarction, or cerebrovascular accident within 6 months prior to study entry.
* History of ventricular rhythm disturbances.
* History of cardiac arrhythmias, stroke, or myocardial infarction.
* Has a cardiac pacemaker.
* History of pericardial effusion or presence of pericardial effusion on screening echocardiogram.
* Taking any medication known to inhibit the cytochrome P450 (CYP)3A4 isozyme or any drugs that are CYP3A4 inducers, or any drugs associated with torsade de pointes or known to prolong the QTcF interval, including anti-arrhythmic medications within 2 weeks prior to screening.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Participant was pregnant, planed to become pregnant, or nursing.
* Human immunodeficiency virus positive.
* Hepatitis B or C positive.
* Immunocompromised.
* Documented renal vascular disease resulting in uncontrolled hypertension.
* Previously received an epithelial growth factor receptor (EGFR).
* Allergy or hypersensitivity to components of tesevatinib or placebo or their formulations.
* Been aphakic due to previous cataract surgery or congenital abnormality.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of California San Diego, La Jolla, California
  - California Institute for Renal Research, La Mesa, California
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale Nephrology Clinical Research, New Haven, Connecticut
  - Coastal Nephrology Associates Research Center, LLC, Port Charlotte, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Rogosin Institute, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 active sites in the United States. A total of 191 participants were screened between 12 October 2017 and 29 January 2020, of which 80 participants were enrolled.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive tesevatinib or placebo.
Groups:
- Tesevatinib: Participants received tesevatinib 50 milligrams (mg) tablet orally once daily (QD) for up to 25.3 months.
Period: Overall Study
Arm/Group | Tesevatinib | Placebo
Started | 40 | 40
Treated | 38 | 40
Completed | 25 | 29
Not Completed | 15 | 11
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Termination of the study by sponsor | 1 | 1
Not completed — Participant moved | 0 | 1
Not completed — Investigator's decision | 3 | 0
Not completed — Other than above specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified Intent-To-Treat (mITT) population which included all randomized participants who receive at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tesevatinib | Placebo | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (9.6) | 45.6 (10.0) | 46.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 14 | 22 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 32 | 33 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Height Adjusted Total Kidney Volume (htTKV) at Month 12
Description: htTKV was calculated using total kidney volume (in milliliters) obtained from magnetic resonance imaging (MRI) divided by height (in meters). Least square (LS) mean and standard error (SE) were estimated by using analysis of covariance (ANCOVA) model. Change from Baseline in htTKV at Month 12 was reported in this outcome measure.
Time Frame: Baseline (Day 1), Month 12
Population: Analysis was performed on efficacy population which included all randomized participants who received at least 1 dose of study drug and completed at least 12 months of tesevatinib or placebo treatment and had a centrally read MRI at Baseline and after 12 months of treatment.
Measure: Least Squares Mean (Standard Error); unit: milliliters per meter
Groups:
- Tesevatinib: Participants received tesevatinib 50 mg tablet orally QD for up to 25.3 months.
Arm/Group | Tesevatinib | Placebo
Number analyzed (Participants) | 31 | 34
milliliters per meter | 0.0236 (0.0059) | 0.0288 (0.0057)
Statistical Analysis 1: Comparison: Tesevatinib vs Placebo; An ANCOVA model included treatment group as a factor and the Baseline htTKV (log10 transformed) as a covariate for the analysis. The outcome measure was tested at 2-sided 0.05 level to control Type I error rate; Test type: Superiority; p = 0.5265, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -0.0052, 95% CI 2-sided [-0.0217 to - 0.0112], Standard Error of Mean 0.0082

2. Primary Outcome: Change From Baseline in Height Adjusted Total Kidney Volume at Month 18
Description: htTKV was calculated using total kidney volume (in milliliters) obtained from MRI divided by height (in meters). LS mean and SE were estimated by using ANCOVA model. Change from Baseline in htTKV at Month 18 was reported in this outcome measure.
Time Frame: Baseline (Day 1), Month 18
Population: Analysis was performed on efficacy population.
Measure: Least Squares Mean (Standard Error); unit: milliliters per meter
Arm/Group | Tesevatinib | Placebo
Number analyzed (Participants) | 31 | 34
milliliters per meter | 0.0383 (0.0081) | 0.0425 (0.0075)
Statistical Analysis 1: Comparison: Tesevatinib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7076, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -0.0042, 95% CI 2-sided [-0.0264 to - 0.0180], Standard Error of Mean 0.0111

3. Primary Outcome: Change From Baseline in Height Adjusted Total Kidney Volume at Month 24
Description: htTKV was calculated using total kidney volume (in milliliters) obtained from MRI divided by height (in meters). LS mean and SE were estimated by using ANCOVA model. Change from Baseline in htTKV at Month 24 was reported in this outcome measure.
Time Frame: Baseline (Day 1), Month 24
Population: Analysis was performed on efficacy population.
Measure: Least Squares Mean (Standard Error); unit: milliliters per meter
Arm/Group | Tesevatinib | Placebo
Number analyzed (Participants) | 31 | 34
milliliters per meter | 0.0485 (0.0103) | 0.0607 (0.0095)
Statistical Analysis 1: Comparison: Tesevatinib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3895, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -0.0122, 95% CI 2-sided [-0.0404 to - 0.0160], Standard Error of Mean 0.0140

4. Primary Outcome: Change From Baseline in Height Adjusted Total Kidney Volume at End of Study
Description: htTKV was calculated using total kidney volume (in milliliters) obtained from MRI divided by height (in meters). LS mean and SE were estimated by using ANCOVA model. Change from Baseline in htTKV at end of study (i.e., up to 26 months) was reported in this outcome measure.
Time Frame: Baseline (Day 1), End of study (anytime up to 26 months)
Population: Analysis was performed on efficacy population.
Measure: Least Squares Mean (Standard Error); unit: milliliters per meter
Arm/Group | Tesevatinib | Placebo
Number analyzed (Participants) | 31 | 34
milliliters per meter | 0.0604 (0.0090) | 0.0589 (0.0094)
Statistical Analysis 1: Comparison: Tesevatinib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9093, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = 0.0015, 95% CI 2-sided [-0.0248 to - 0.0278], Standard Error of Mean 0.0131

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal product and which did not necessarily had to have a causal relationship with the treatment. TEAEs were AEs that developed or worsened or became serious from the first dose (Day 1) of the study drug until end of study.
Time Frame: From Baseline (Day 1) up to 30 days post last dose of study drug (i.e., up to 26 months)
Population: Analysis was performed on safety population which included all participants who received at least 1 dose of study drug and were analyzed according to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Tesevatinib | Placebo
Number analyzed (Participants) | 38 | 40
Participants | 37 | 40

6. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Months 12, 18, 24 and End of Study
Description: eGFR is a test for renal function. eGFR was calculated by using the 4-variable modification of diet in renal disease (MDRD-4) formula reported as milliliters per minute per 1.73 square meter (mL/min/1.73 m^2). LS mean and SE were estimated using ANCOVA model.
Time Frame: Baseline (Day 1), Months 12, 18, 24 and at end of study (i.e., anytime up to 26 months)
Population: Analysis was performed on efficacy population.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Tesevatinib | Placebo
Number analyzed (Participants) | 31 | 34
mL/min/1.73m^2
  Month 12 | -6.8032 (1.2293) | -2.1780 (1.1709)
  Month 18 | -7.3626 (1.6645) | -3.8950 (1.6971)
  Month 24 | -9.7307 (1.4708) | -6.4070 (1.4138)
  End of study | -3.2757 (0.5990) | -3.7497 (0.6323)

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) up to 30 days post last dose of the study drug (i.e., up to 26 months)
Description: Reported AEs were TEAEs that developed or worsened or became serious from the first dose (Day 1) of the study drug up to end of the study. Analysis was performed on safety population.
Arm/Group | Tesevatinib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 6/38 | 2/40
Other Adverse Events (participants affected / at risk) | 37/38 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tesevatinib (N=38) | Placebo (N=40)
Appendicitis (Infections and infestations) | 0 | 1
Renal cyst infection (Infections and infestations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tesevatinib (N=38) | Placebo (N=40)
Diarrhoea (Gastrointestinal disorders) | 21 | 13
Nausea (Gastrointestinal disorders) | 14 | 6
Vomiting (Gastrointestinal disorders) | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 5
Abdominal discomfort (Gastrointestinal disorders) | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 12 | 12
Upper respiratory tract infection (Infections and infestations) | 7 | 6
Urinary tract infection (Infections and infestations) | 5 | 4
Gastroenteritis viral (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Otitis media (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 9 | 6
Acne (Skin and subcutaneous tissue disorders) | 6 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 13 | 9
Dizziness (Nervous system disorders) | 12 | 0
Paraesthesia (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 6
Amylase increased (Investigations) | 4 | 2
Alanine aminotransferase increased (Investigations) | 1 | 4
Blood creatinine increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 4
Blood potassium increased (Investigations) | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 3 | 0
Blood bicarbonate decreased (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 2 | 0
Oedema peripheral (General disorders) | 2 | 6
Pyrexia (General disorders) | 2 | 4
Fatigue (General disorders) | 1 | 4
Chills (General disorders) | 1 | 3
Pain (General disorders) | 0 | 4
Oedema (General disorders) | 1 | 2
Peripheral swelling (General disorders) | 1 | 2
Influenza like illness (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 3 | 4
Renal pain (Renal and urinary disorders) | 2 | 5
Renal cyst ruptured (Renal and urinary disorders) | 1 | 3
Dysuria (Renal and urinary disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 1
Vision blurred (Eye disorders) | 3 | 1
Dry eye (Eye disorders) | 1 | 2
Ocular hyperaemia (Eye disorders) | 2 | 0
Optic nerve disorder (Eye disorders) | 0 | 2
Photophobia (Eye disorders) | 2 | 0
Retinal haemorrhage (Eye disorders) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Muscle strain (Injury, poisoning and procedural complications) | 2 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 2
Hypertension (Vascular disorders) | 4 | 4
Hypotension (Vascular disorders) | 1 | 2
Flushing (Vascular disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cyst (Reproductive system and breast disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03203642/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT03203642/SAP_001.pdf